CLINICAL TRIAL: NCT04847193
Title: Effect of Iso-alpha-Acids and Xanthohumol on Inflammatory Processes in Human
Brief Title: Hop Compounds and Immune System
Acronym: HI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ina Bergheim, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UVienna19a
Record Dates: First submitted 2021-03-16; First posted 2021-04-19 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Inflammatory Response

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Experimental): Participants receive a study drink supplemented with a placebo over a time period of 5 days.
  Interventions: Other: Dietary Intervention 1: Placebo
- Xanthohumol (Experimental): Participants receive a study drink supplemented with Xanthohumol over a time period of 5 days.
  Interventions: Other: Dietary Intervention 2: Xanthohumol and Iso-alpha acids
- Iso-alpha acids (Experimental): Participants receive a study drink supplemented with Iso-alpha acids over a time period of 5 days.
  Interventions: Other: Dietary Intervention 2: Xanthohumol and Iso-alpha acids
- Xanthohumol/Iso-alpha acids (Experimental): Participants receive a study drink supplemented with a combination of Xanthohumol and Iso-alpha acids over a time period of 5 days.
  Interventions: Other: Dietary Intervention 2: Xanthohumol and Iso-alpha acids

INTERVENTIONS:
Other: Dietary Intervention 1: Placebo — Participants receive a study drink supplemented with a placebo for 5 days
  Arms: Placebo
Other: Dietary Intervention 2: Xanthohumol and Iso-alpha acids — Participants receive a study drink supplemented with xanthohumol, Iso-alpha acids or a combination of both for 5 days
  Arms: Iso-alpha acids; Xanthohumol; Xanthohumol/Iso-alpha acids

SUMMARY:
The aim of the present study is to determine the effect of Xanthohumol and Iso-alpha-acids from hops on the immune response of healthy participants.

DETAILED DESCRIPTION:
In this placebo-controlled crossover study a study drink enriched with either a placebo, Xanthohumol, Iso-alpha Acids or a combination of latter is given to the participants. A washout phase before intervention and between each intervention is introduced. On day one of each intervention blood is drawn in fasted state from each participant. Subsequently the study drink combined with a standardized breakfast is given to the participants following a second blood drawing one hour after the consumption of the study drink. On the last day of each intervention blood is taken from study participants in the same manner as on day one. To assess the effect of Xanthohumol and Iso-alpha acids or a combination of both, clinical chemical parameters e.g. ALT, AST, γ-GT, blood lipids (triglycerides, total cholesterol, HDL, LDL), blood glucose, uric acid and CRP are determined. Furthermore, PBMC's isolated from blood samples of each time point were stimulated for either 24 or 48 h. Protein levels and mRNA expression of markers of inflammation is measured in PBMC's and supernatant of stimulated cells.

ELIGIBILITY:
Inclusion Criteria:

* healthy, normal weight,

Exclusion Criteria:

* food intolerances, food allergies, chronic inflammatory diseases, metabolic diseases, viral or bacterial infections within the last 3 weeks of inclusion, intake of immunosupressive medication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Changes in parameters of immune response | 5 days
  Parameters of immune response are measured in cell culture supernatant of stimulated cells

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung F, Staltner R, Baumann A, Burger K, Halilbasic E, Hellerbrand C, Bergheim I. A Xanthohumol-Rich Hop Extract Diminishes Endotoxin-Induced Activation of TLR4 Signaling in Human Peripheral Blood Mononuclear Cells: A Study in Healthy Women. Int J Mol Sci. 2022 Oct 21;23(20):12702. doi: 10.3390/ijms232012702. PMID 36293555
- [Derived] Jung F, Staltner R, Tahir A, Baumann A, Burger K, Halilbasic E, Hellerbrand C, Bergheim I. Oral intake of xanthohumol attenuates lipoteichoic acid-induced inflammatory response in human PBMCs. Eur J Nutr. 2022 Dec;61(8):4155-4166. doi: 10.1007/s00394-022-02964-2. Epub 2022 Jul 20. PMID 35857130